CLINICAL TRIAL: NCT02213939
Title: Removal of Cytokine on Cardiopulmonary Bypass With CytoSorb® Compared to on- and Off-pump Myocardial Revascularization
Brief Title: Clinical Impact of Cytokine in Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Antje-Christin Deppe, MD, Resident Cardiac Surgery, University Hospital of Cologne
Other Study IDs: Cytosorb2014
Record Dates: First submitted 2014-08-04; First posted 2014-08-12 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Coronary Disease
Keywords: Myocardial revascularization; Cytosorb; Inflammatory response; Cardiopulmonary bypass
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- CPB + Cytosorb: On pump myocardial revascularization with the use of the cytokine adsorbing circuit (Cytosorb)
- CPB / Control: Controll group; on pump myocardial revascularization
- OPCAB / Control: Controll Group; off-pump myocardial revascularization

SUMMARY:
Cardiac surgery leeds to a systematic inflammatory response induced by the surgical trauma and the use of the cardiopulmonary bypass (CPB). Activation of inflammatory cascades can cause a systemic inflammatory response syndrome (SIRS) which is associated with increased morbidity and mortality. Therefore, strategies to reduce the inflammatory response have a potential benefit for cardiac surgery patients.

The clinical benefit of reducing proinflammatory cytokines such as IL-6, Il-8 and TNF-a with the use of a cytokine adsorbing circuit (Cytosorb) during CBP remains unclear. Therefore, the investigators conduct this prospective, observational pilot study to determine the clinical impact of the use of a cytokine adsorbing circuit during CBP.

DETAILED DESCRIPTION:
Patients, who have an elective myocardial revascularization and give there written consent will be enrolled to the study. Demographic, intraoperative, and postoperative data will be collected prospectively. Furthermore, blood samples (1. before induction of anaesthesia 2. at the end of CPB 3. 6 hours after surgery 4. 24 hours after surgery 5. 3-5 days after surgery) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* • Elective myocardial revascularization

Exclusion Criteria:

* Emergency procedures
* Declined informed consent
* Body mass index < 18
* Age < 18 years
* Pregnant women
* Receiving chemotherapy
* Diagnosed with any disease state (e.g., AIDS) that has produced leukopenia
* Receiving antileukocyte drugs
* Receiving TNF-α Blockers
* Receiving immunosuppressive drugs or hormone therapy (e.g. tamoxifen)
* CRP > 5 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving surgical myocardila revascularization
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Evolution of the inflammatory response | Change from Baseline in cytokine level direct after surgery, 6 and 24 hours after surgery; 5. postoperative day
  Il-6; Il-8; TNF-a; C3/C4-complement Leucocytes CRP

SECONDARY OUTCOMES:
Length of ICU and hospital stay | participants will be followed for the duration of hospital stay, an expected average of 10 days
  Length of ICU and hospital stay
Length of ventilation | participants will be followed for the duration of hospital stay, an expected average of 10 days
  Length of ventilation (hours)
Length of catecholamine therapy | participants will be followed for the duration of hospital stay, an expected average of 10 days
  Length of catecholamine therapy
kidney injury | participants will be followed for the duration of hospital stay, an expected average of 10 days
  kidney injury defined as an increase in SCr by ≥1.0 mg/dl (≥26.5 μmol/l) after surgery ; or Increase in SCr to ≥1.5 times baseline, or Urine volume < 0.5 ml/kg/h for 6 hours.
MACCE (mortality; myocardial infarction; cerebrovascular accident) | participants will be followed for the duration of hospital stay, an expected average of 10 days
  Mortality measured as any kind of death and myocardial death Myocardial Infarction measured with ECG; CK-MB, cTnT Cerebrovascular accident verified with abnormal cerebral CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Antje C Deppe, MD, Principal Investigator — University Hospital of Cologne; Department of Cardiothoracic Surgery;
Locations (1):
- University Hospital of Cologne; Department of Cardiothoracic Surgery, Cologne, Germany